CLINICAL TRIAL: NCT05938270
Title: An Open-label, Randomised, Phase-I, Multi-Centre Study to Investigate the Biological Effects of Saruparib (AZD5305) Alone, Darolutamide Alone, and in Combination Given Prior to Radical Prostatectomy in Men With Newly Diagnosed Prostate Cancer (ASCERTAIN)
Brief Title: A Study to Investigate the Biological Effects of Saruparib (AZD5305), Darolutamide, and in Combination in Men With Newly Diagnosed Prostate Cancer.
Acronym: ASCERTAIN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D9721C00002; 2023-503691-25-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-05-16; First posted 2023-07-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer, radical prostatectomy, Darolutamide, Saruparib (AZD5305)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — AZD5305; darolutamide

STUDY DESIGN:
Intervention Model Description: Randomised, phase 1 multicentre study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Saruparib (AZD5305) only (Other): Participant will receive Saruparib (AZD5305) once daily for 21 days (+ up to 7 days) unless unacceptable toxicity or withdrawal of consent. Following the 21 days of study treatment, participants should undergo radical prostatectomy on Day 22 (+ up to 7 days)
  Interventions: Drug: Saruparib (AZD5305)
- Saruparib (AZD5305) + Darolutamide (Other): Participant will receive Saruparib (AZD5305) once daily + darolutamide twice daily for 21 days (+ up to 7 days) unless unacceptable toxicity or withdrawal of consent. Following the 21 days of study treatment, participants should undergo radical prostatectomy on Day 22 (+ up to 7 days).
  Interventions: Drug: Saruparib (AZD5305); Drug: Darolutamide
- No Treatment (Other): No study treatment is to be taken by the participants in this arm. Radical prostatectomy should be performed as per local practice
  Interventions: Other: No Treatment
- Darolutamide Only (Other): Participant will receive darolutamide twice daily for 21 days (+ up to 7 days) unless unacceptable toxicity or withdrawal of consent. Following the 21 days of study treatment, participants should undergo radical prostatectomy on Day 22 (+ up to 7 days).
  Interventions: Drug: Darolutamide

INTERVENTIONS:
Drug: Saruparib (AZD5305) — Saruparib (AZD5305) given orally once daily
  Other Names: Darolutamide is also known as Nubeqa
  Arms: Saruparib (AZD5305) + Darolutamide; Saruparib (AZD5305) only
Drug: Darolutamide — Darolutamide tablet is 300mg, given BD orally, twice daily- total dose 1200mg
  Other Names: Darolutamide is also known as Nubeqa
  Arms: Darolutamide Only; Saruparib (AZD5305) + Darolutamide
Other: No Treatment — No study treatment is to be taken by the participants in this arm. Radical prostatectomy should be performed as per local practice
  Arms: No Treatment

SUMMARY:
A Study to Investigate the Biological Effects of Saruparib (AZD5305) Alone, Darolutamide Alone, and in Combination Given Prior to Radical Prostatectomy in Men with Newly Diagnosed Prostate Cancer (ASCERTAIN).

DETAILED DESCRIPTION:
An Open-label, Randomised, Phase-I, Multi-Centre Study to Investigate the Biological Effects of Saruparib (AZD5305) alone, Darolutamide alone, and in Combination Given Prior to Radical Prostatectomy in Men with Newly Diagnosed Prostate Cancer (ASCERTAIN).

ELIGIBILITY:
Inclusion Criteria:

* male participants >/= 18 years old
* participants deemed suitable for radical prostatectomy
* participants with localised prostate cancer with unfavourable intermediate/high/very high risk eligible for prostatectomy
* adequate organ and marrow function as per protocol
* capable of giving signed informed consent
* For participants participating in the Optional Genetic Research Only: Provision of signed and dated written Optional Genetic Research Information
* Available FFPE diagnostic tumour biopsy samples
* Participants must use a condom (with spermicide) from screening to 6 months after screening and refrain from fathering a child or donating sperm

Exclusion Criteria:

* As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including, active bleeding diatheses, or active infection including HepB, hepatitis C and HIV. Screening for chronic conditions is not required.

  1. Active HBV is defined by a known positive HBsAg result. Participants with a past or resolved HBV infection (defined as the presence of HepB antibody and absence of HBsAg) are eligible.
  2. Participants positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Participants with any known predisposition to bleeding (eg, active peptic ulceration, recent [within 6 months] haemorrhagic stroke, proliferative diabetic retinopathy).
* Participants with history of MDS/AML or with features suggestive of MDS/AML (as determined by prior diagnostic investigation). In case there is no Clinical MDS/AML suspicion, no specific screening for MDS/AML (by bone marrow/bone biopsy) is required.
* Prior malignancy within 3 years of screening whose natural history, in the Investigator's opinion, has the potential to interfere with safety and efficacy assessments of the investigational regimen.
* Concomitant use of drugs that are known to prolong or shorten QT and have a known risk of TdP.
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTcF) > 450 milliseconds or QTcF < 340 milliseconds obtained from triplicate ECGs and averaged, recorded within 5 minutes.
  2. Any factors that increase the risk of QT prolongation, shortening or risk of arrhythmic events such as hypokalaemia, congenital long or short QT syndrome, family history of long QT syndrome, familial short QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong or shorten the QT interval.
  3. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, second or third degree atrioventricular block and clinically significant sinus node dysfunction not treated with pacemaker.
* Other CVS diseases as defined by any of the following:

  1. Symptomatic heart failure (as defined by NYHA class ≥ 2).
  2. uncontrolled hypertension.
  3. hypertensive heart disease with significant left ventricular hypertrophy.
  4. History of acute coronary syndrome/acute myocardial infarction, unstable angina pectoris, coronary intervention procedure with percutaneous coronary intervention or coronary artery bypass grafting within 6 months prior to screening.
  5. cardiomyopathy of any aetiology.
  6. presence of clinically significant valvular heart disease.
  7. history of atrial or ventricular arrhythmia requiring acute treatment; participants with atrial fibrillation and optimally controlled ventricular rate (heart rate < 100 bpm) are permitted.
  8. transient ischaemic attack, or stroke within 6 months prior to screening.
  9. participants with symptomatic hypotension at screening.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of Saruparib (AZD5305).
* History of prior malignancy, treated with chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, or other anticancer agent within 3 years of screening. Previously localised surgically treated malignancy is acceptable, if no evidence of recurrence.
* Known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s).
* Prior treatment with any systemic or localised anti-cancer treatment for the localised prostate cancer.
* During the 4 weeks prior to the first dose, receiving immune modulatory agents including but not limited to, continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent.
* Concomitant use of medications or herbal supplements known to be:

  1. Strong CYP3A4 inducers/inhibitors (applies for Saruparib (AZD5305) and Saruparib (AZD5305) + darolutamide arms)
  2. Strong or moderate CYP3A4 and P-glycoprotein inducers (applies to darolutamide arm and Saruparib (AZD5305) + darolutamide arm) This is including, but not limited to, the prohibited medications listed in CSP Appendix G, or inability to stop the use thereof, at least 21 days or at least 5 half-lives (whichever is longer) before the first dose of study treatment until 30 days after the last dose of study treatment.
* Treatment with any investigational agents or study interventions from a previous clinical study within 5 half-lives or 3 weeks (whichever is longer) of the first dose of study treatment.
* Participants with contraindication to darolutamide for treatment arms
* Unable to comply with the visits and assessments.
* In the opinion of the Investigators should not be included in this study.

No treatment arm only: if any participant meets exclusion 4, 9 or 11, they are not to be included in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants >/=18 years of age
Enrollment: 120 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-08-17 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Fold change in % γH2AX positive cells from baseline value in tumour samples | Tumour biopsy taken at diagnosis within approx 2 months of Day 1 planned start of study treatment; post treatment tumour biopsy taken following 21 days (+ up to 7 days) of study treatment
  To assess the effects of study treatment on γH2AX change in participants with localised prostate cancer

SECONDARY OUTCOMES:
Severity of Treatment-Emergent AEs/SAEs per CTCAE v5.0 | Day 1 to 28 days post-surgery
  To assess the safety and tolerability of study treatment in participants with localised prostate cancer
Incidence of Treatment-Emergent AEs/SAEs per CTCAE v5.0 | Day 1 to 28 days post-surgery
  To assess the safety and tolerability of study treatment in participants with localised prostate cancer
Number of patients with abnormal laboratory values | Day 1 to 28 days post-surgery
  To assess the safety and tolerability of study treatment in participants with localised prostate cancer
Change from baseline in blood pressure reported as clinically significant | Day 1 to 28 days post-surgery
  To assess the safety of study treatment in participants with localised prostate cancer
Change from baseline in heart rate reported as clinically significant | Day 1 to 28 days post-surgery
  To assess the safety of study treatment in participants with localised prostate cancer
Change from baseline in QTc value | Day 1 to 28 days post-surgery
  To assess the safety of study treatment in participants with localised prostate cancer
Number of participants undergoing planned surgery | Measured based on Day 1 to Day 21 of treatment
  To assess the impact of study treatment on surgical feasibility in participants with localised prostate cancer
Reasons of participants requiring treatment-related and non-treatment related delays of surgery and delays > 7 days from scheduled day | Measured based on Day 1 to Day 21 of treatment
  To assess the impact of study treatment on surgical feasibility in participants with localised prostate cancer
Number of participants requiring treatment-related and non-treatment related delays of surgery and delays > 7 days from scheduled day | Measured based on Day 1 to Day 21 of treatment
  To assess the impact of study treatment on surgical feasibility in participants with localised prostate cancer
Change in Ki-67 % positive cells from baseline in tumour samples | Measured based on Day 1 to Day 21 of treatment
  To assess the effects of study treatment on Ki-67 change in participants with localised prostate cancer

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - Research Site, Detroit, Michigan
  - Research Site, Providence, Rhode Island
- Australia (2):
  - Research Site, Melbourne
  - Research Site, South Brisbane
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Valencia
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Istanbul
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home